CLINICAL TRIAL: NCT02538211
Title: The Role of the Intestinal Microbiome in Enteric and Systemic Vaccine Immune Responses
Acronym: Rota-biome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Wageningen University and Research (Other)
Responsible Party: Principal Investigator, W.J. Wiersinga, MD, PhD, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL 52510.018.15
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Rotavirus Infections; Intestinal Bacteria Flora Disturbance; Reaction - Vaccine Nos; Tetanus; Streptococcal Pneumonia
MeSH Terms: conditions — Rotavirus Infections; Tetanus; Pneumonia | interventions — Rotavirus Vaccines; Tetanus Toxoid; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Control group - subjects will receive no antibiotics
  followed by Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine
  Interventions: Biological: Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine
- Broad-spectrum antibiotics (Active Comparator): Subjects will receive 7 days of pre-treatment (days -9 to -3) with:
  * Ciprofloxacin 500mg 2dd1
  * Vancomycin 250mg 3dd2
  * Metronidazole 500mg 3dd1
  followed by Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine
  Interventions: Biological: Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine
- Narrow-spectrum antibiotics (Active Comparator): Subjects will receive 7 days of pre-treatment (days -9 to -3) with:
  • Vancomycine 250mg 3dd2
  followed by Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine
  Interventions: Biological: Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine

INTERVENTIONS:
Biological: Rotavirus vaccine, Tetanus vaccine and Pneumococcal vaccine — All subjects will be given an oral dose of the rotavirus vaccine, RotarixTM, and intramuscular injections of the Tetanus vaccine and Pneumococcal vaccine, Pneumo 23.
  Other Names: RotarixTM, Pneumo 23

SUMMARY:
The purpose of this study is to evaluate if the intestinal microbiota influences rotavirus vaccine immune responses in healthy adult volunteers.

DETAILED DESCRIPTION:
This study will alter the intestinal microbiota in healthy adults using antibiotics and subsequently measure immune reactions to the rotavirus vaccine (Rotarix), the tetanus vaccine and the pneumococcal vaccine (Pneumo23).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible physician, based on a medical evaluation including medical history, physical examination and laboratory tests carried out within 28 days prior to starting antibiotics (day -98). A subject with a clinical abnormality or laboratory parameter outside the reference range may be included if the investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male between 18 and 35 years of age, inclusive at the time of signing the informed consent
* Capable of giving written informed consent and able to comply with the requirements and restrictions listed in the informed consent form
* Normal defecation pattern (defined as ≤3x/ day and ≥3x/week)

Exclusion Criteria:

* Subject has had a major illness in the past 3 months or any significant chronic medical illness that the investigator would deem unfavorable for enrollment, including inflammatory diseases.
* Subject with any history of immunodeficiency
* Subjects with a history of any type of malignancy
* Subject with a history of thrombocytopenia or bleeding disorder
* Subject has a past or current gastrointestinal disease which may influence the gut microbiota
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of alcoholism and/or drinking more than an average of 5 units of alcohol per day
* The subject has received an investigational product within three months of day 0 of the current study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Height of serum anti-rotavirus Immunoglobulin A (IgA) response | 28 days post-vaccination
  Geometric Mean Concentration (GMC)

SECONDARY OUTCOMES:
Time to positivity for serum anti-rotavirus Immunoglobulin A (IgA) and G (IgG) response | day 0 through day 28 post vaccination
  (days)
Change in pre and post-vaccination anti-rotavirus (anti-RV) serum neutralizing antibodies measured by Geometric Mean Concentration (GMC) | 28 days post-vaccination
Change in pre and post-vaccination anti-RV serum IgG response measured by Geometric Mean Concentration (GMC) | day 0 through day 28 post vaccination
Change in serum tetanus toxoid IgG response, measured as pre and post vaccination titer (international units/mL) ratio | day 0 through day 28 post vaccination
Change in serum pneumococcal poly-saccharide-specific IgG for all vaccine strains , measure in pre and post vaccination titer (micrograms/mL) ratio | day 0 through day 28 post vaccination
Composition of the fecal micro biome before and after antibiotics and between groups measured by the HITChip and bacterial 16S rRNA sequencing | day -9 and day 0 pre vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Willem J. Wiersinga, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands